CLINICAL TRIAL: NCT04257266
Title: The Effect of 5-site Ice Pack Cooling on Body Temperature, Skin Temperature, and Heart Rate After Exercise-induced Hyperthermia
Brief Title: Cryo Pack Cooling After Exercise-induced Hyperthermia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding was never received and the study was terminated in the IRB
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Douglas J Casa, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H19-168
Record Dates: First submitted 2019-12-10; First posted 2020-02-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Participants receive two alternative interventions: 1) cryothermic cooling pack and 2) commercially available ice pack.
Who Masked: Participant
Masking Description: The participant will be blinded to which ice pack will be used during the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryo Cooling Pack (Experimental): Cryo cooling pack will be placed on subjects for 30 mins after exercise-induced hyperthermia is achieved.
  Interventions: Device: Ice Pack Cooling
- Commerical Ice Pack (Active Comparator): The commercial ice pack will be placed on subjects for 30 mins after exercise-induced hyperthermia is achieved.
  Interventions: Device: Ice Pack Cooling

INTERVENTIONS:
Device: Ice Pack Cooling — 5 ice packs (Cryo cooling pack or commercial ice pack) will be placed on the subject for 30 mins after exercise-induced hyperthermia

SUMMARY:
This research study aims to examine whether Cryo Cooling packs reduce thermal and cardiovascular strain after exercise-induced hyperthermia compared to a commercially available ice pack. Secondly, the effect of Cryo Cooling packs on cognitive and exercise performance will be examined. There is no current research examining the efficacy of Cryo Cooling packs in hyperthermic individuals and this information will be helpful to establish whether Cryo Cooling Packs can be used for performance enhancement or to prevent heat illness.

DETAILED DESCRIPTION:
This study will consist of three study visits:

Visit 1: Baseline and VO2max Testing Visit 2-3: Trial 1 and 2.

Visit 1: Baseline and VO2max Testing

Participants who are approved to participate will be scheduled for a baseline and VO2max testing day. Upon arrival to the lab, subjects will provide a urine sample in a clean urine cup. Urine specific gravity and urine color will be assessed. Nude body mass will be also be recorded. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room behind a solid, closed door, and the research reading the scale outside of the room. Participants will only be permitted to continue to the VO2max test if the euhydrated criteria of a urine specific gravity (USG) ≤1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status. Height will be measured with a tape measure on Visit 1. Percent body fat will be calculated using a 3-site evaluation of skin fold thickness using skin fold calipers on one of the three baseline days. A researcher will use appropriate grasping technique to measure skin fold thickness on the chest, abdomen, and thigh. This will take less than ~5 minutes to complete. This information will be used to describe the subject demographics. Participants will also be asked to complete a maximal oxygen uptake (VO2max) test on a treadmill in a thermoneutral environment. This test will provide aerobic fitness levels of the participants.

Visit 2-3: Trials 1 and 2

This is a randomized, counter-balanced, cross over design. Participant numbers will be randomly assigned and trials will be ordered with a random number generator and assigned to a participant number. These orders will be counterbalanced between participants to ensure that there is not an order effect, and each participant will complete both trials as part of the study. Participants will be allowed to make-up trial visits if they are sick, suffer an injury or do not meet hydration requirements. Participants will be asked if they have a current illness or taking medications to determine whether they can complete the exercise trial. The participant's visit will be rescheduled if they have a fever, current illness or taking medications that influence body temperature.

Cooling Intervention:

1. Ice Pack Cooling
2. Commercially Available Ice Pack

The exercise protocol, performance testing, cognitive testing, and recovery portions of this study will be conducted in a climatic chamber with ambient temperature approximately 30-40°C and relative humidity at approximately 30-70%.

Upon arrival to the lab, participants will be asked to indicate if they have consumed alcohol or caffeine in the last 24 hours. They will not be asked to specify exactly what they have consumed, but if they provide a positive indication, their trial will be rescheduled for another day. Participants will provide a small urine sample in a clean urine cup, and a nude body mass will be measured. Upon arrival to the lab, hydration status will be assessed by urine specific gravity, nude body mass and urine color. Participants will only be permitted to continue to the exercise trial if the euhydrated criteria of a urine specific gravity (USG) ≤ 1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status. Participants will be given instructions at the prior visit about how to obtain desired hydration status for the upcoming trial. Key study personnel will insert an esophageal probe to measure esophageal temperature. Participants will then insert a rectal probe and wear a heart rate monitor strap. Additionally, participants will wear 4-site skin temperature sensors. The participants will also be asked to complete a subjective sleep questionnaire upon arriving to the lab. All perceptual measures, cognitive performance measures and physical performance tests will be administered to determine a baseline value at the beginning of each trial.

All participants will undergo a treadmill protocol involving approximately 90 minutes of jogging or walking. Cognitive and physical performance tests will be administered at various time points throughout the trial.

After exercise, participants will be cooled by either 5 cryothermic ice packs or 5 commercially available ice packs. Participants will be cooled for approximately 30 mins. All participants will be laying supine during cooling.

Cryothermic Cooling and Commercially Available Ice Pack Placement

Storage and Preparation:

Ice packs will be stored in a cooler at approximately 34°F for at least 6 hours prior to use and kept as dry as possible (35°F to 70°F). Ideally, Ice packs will be kept in tray or basket above ice or frozen gel packs, not in contact with the method of cooling the cooler. Refrigerator may be acceptable for storage before cooler use as well, but prefer cooler for real situations in field.

For cryo cooling elements: the cryo cooling packs will be shaken quickly and vigorously (10 seconds) and placed on subject (subject will be supine).

For commercially available ice pack: ice packs will be placed on subject (subject will be supine).

All ice packs will be placed on the following body segments:

* 1 ice pack on neck covering both carotid Triangle regions
* 2 ice packs in axilla region
* 2 ice packs in groin region

Cryo Cooling Elements and commercially available ice packs will be discarded after use.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30 years
* been cleared by the medical monitor for this study

Exclusion Criteria:

* Have a current musculoskeletal injury that would limit their physical activity or preclude the participant from walking, jogging, running, sprinting, or cutting.
* Chronic health problems that affect your ability to thermoregulate (disorders affecting the liver, kidneys or the ability to sweat normally)
* Fever or current illness at the time of testing
* History of cardiovascular, metabolic, or respiratory disease
* Current musculoskeletal injury that limits their physical activity
* Currently taking a medication that is known to influence body temperature (amphetamines, antihypertensives, anticholinergics, acetaminophen, diuretics, NSAIDs, aspirin)
* Are a female
* Have a history of heat related illness
* Throat or gastroesophageal diseases including gastroesophageal reflux disease (aka, GERD) or difficulty swallowing

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Rectal Temperature | Measured continuously for 2-3 hours during exercise and cooling period
  Rectal thermometer will be self-inserted by participant to assess core temperature
Change in Esophageal Temperature | Measured continuously for 2-3 hours during exercise and cooling period
  Esophageal thermometer will be inserted by trained personnel to assess core temperature
Change in Heart rate | Measured continuously for 2-3 hours during exercise and cooling period
  A heart rate monitor will be worn by participant throughout exercise/cooling protocol
Change in Skin Temperature | Measured continuously for 2-3 hours during exercise and cooling period
  4 skin temperature sensors will be placed on the subject (chest, shoulder, thigh, calf) during exercise and the cooling intervention
Change in Rating of Perceived Exertion | Collected every 5 minutes during 2-3 hour exercise and cool down period.
  6-20 scale that indicates how hard the participant feels they are working
Change in Perception of Fatigue | Collected every 5 minutes during 2-3 hour exercise and cool down period.
  0-10 (no fatigue to extreme fatigue) Scale that indicates how fatigued the participate feels
Change in Perception of Thirst | Collected every 5 minutes during 2-3 hour exercise and cool down period.
  0-9 (no thirst to very,very thirsty) Scale that indicates how thirsty the participant is
Change in Thermal Sensation | Collected every 5 minutes during 2-3 hour exercise and cool down period.
  0-8 Scale (cold to hot) that indicated how cold or hot the participate feels

SECONDARY OUTCOMES:
Profile of Mood States | Immediately before exercise
  Questionnaire that indicates the current mood of the participant
Profile of Mood States | immediately following exercise
  Questionnaire that indicates the current mood of the participant
Profile of Mood States | immediately following cooling intervention
  Questionnaire that indicates the current mood of the participant
Reaction time test | immediately before exercise
  A ruler drop test to test reaction time
Reaction time test | immediately after exercise
  A ruler drop test to test reaction time
Reaction time test | immediately after cooling intervention
  A ruler drop test to test reaction time
Digits Backwards | immediately before exercise
  A test where participants are asked to repeat digits backwards to examine memory
Digits Backwards | immediately after exercise
  A test where participants are asked to repeat digits backwards to examine memory
Digits Backwards | immediately after cooling intervention
  A test where participants are asked to repeat digits backwards to examine memory
1 Mile run | immediately following Cooling
  A treadmill test where participants run as fast they can for 1 mile
Grip strength: Hand Grip Dynamometer | immediately following cooling
  Participant will squeeze a hand drip dynamometer (one hand at a time) for 3 trials to estimate grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Casa, PhD, Principal Investigator — University of Connecticut

IPD SHARING:
Plan to Share IPD: No
Analyzed and summary data will be shared through publication in a journal article